CLINICAL TRIAL: NCT01358838
Title: Ablative 10600 nm Fractional Laser Therapy for the Treatment of Scars; a Randomized Controlled Trial
Brief Title: Ablative 10600 nm Fractional Laser Therapy for the Treatment of Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Netherlands Institute for Pigment Disorders, Netherlands Institute for Pigment Disorders
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC 10/026
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2010-05

CONDITIONS: Scars
Keywords: Patients with either hypertrophic or atrophic scars; Efficacy of ablative 10600nm fractional laser therapy; Laser therapy compared to no treatment of (part of) the scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- laser (Active Comparator)
  Interventions: Device: ablative 10600 nm fractional laser therapy
- no laser (No Intervention)

INTERVENTIONS:
Device: ablative 10600 nm fractional laser therapy — Half of the scar, or one of two comparable scars, will be treated with the ablative 10600 nm fractional laser. There wil be 3 treatments, with 8 weeks apart.
  Half of the scar, or one of two comparable scars, will receive no treatment at all.
  Arms: laser

SUMMARY:
Rationale: Scars can be highly disfiguring and may result in functional impairment and psychosocial problems. Recently, fractional laser therapy (FLT) has been introduced as a promising novel treatment modality for scars.

Objectives: The primary objective of this study is to assess the efficacy and safety of 10600 nm FLT for the treatment of different types of scars.

Study design: Prospective observer blinded randomised controlled split-lesion trial.

Study population: Thirty consecutive patients, aged at least 18 years, with hypertrophic or atrophic scars who give written informed consent.

Methods: Two similar test regions of the scar will be randomly allocated to either 3 sessions of FLT (UltraPulse Encore 10600 nm Total FX) with an interval of 4 weeks or no treatment.

Main study parameters/endpoints: Blinded Physicians Global Assessment is the main outcome variable. Secondary variables are Patient's Global Assessment, blinded clinical assessment of the scar on a scale from 0-3 (erythema, pigmentation, texture, hypertrophy, atrophy, pliability), Patient and Observer Scar Scale (POSAS), objective colour measurements by reflectance spectroscopy (LAB) and chromameter (erythema index, melanin index).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects participating in the study will be requested to visit the SNIP (Amsterdam) 3 times for treatment and 2 times for follow-up. The time investment per visit will be 30 minutes for treatment sessions and 20 minutes for follow-up visits. FLT using a 10600 nm laser device is a minimally invasive laser procedure with FDA approval for both the device (Lumenis Encore 10600 nm) and the indication (scar). Local side effects are erythema (always; 1-2 weeks), oozing (often; 1-3 days), swelling (always, 1-4 days), blisters < 0.5cm (occasionally) and blisters > 0.5cm (very rare). No systemic side effects are known for this laser device.

All outcome measures involve non-invasive procedures. The laser treatment (FLT) requires local anesthesia. The amount of topical anesthetic used for infiltration is low (approximately 5% of the maximum dose) which minimizes the risk for local or systemic side effects due to the anesthetic agent.

All together the burden due to the study is moderate, side effects are generally local and mild. Systemic side effects are not reported with this treatment. There is an indirect benefit for the participating subject. In case of improvement of the treated test regions, this therapy can be directly utilized to treat the whole scar.

Considering the relative lack of alternative treatment options in many of these scars, the balance between burden, possible side effects and prospect for improvement is very favorable.

ELIGIBILITY:
Inclusion Criteria:

* Atrophic or hypertrophic scars allowing for demarcation of two similar test regions of at least 2x2cm
* Age at least 18 years
* Subject is willing and able to give written informed consent
* Interval between injury and start of study at least one year

Exclusion Criteria:

* Suspected allergy to lidocaine
* Use of roaccutane (isotretinoin) in the past 12 months
* Subjects not competent to understand what is involved
* Skin type V and VI
* Pregnancy
* Concomitant skin disease at the site of treatment
* Presence of lesions suspicious for malignancy in the scar
* High exposure to sunlight (vacation in southern countries) or UV light (UVA or UVB) during the first 4 weeks after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement of the scar | 18 months
  Improvement of erythema, pigment, and structure of the scar assessed by a blinded dermatologist (blinded physician global assessment) and by objective colour measurements (chromameter)

SECONDARY OUTCOMES:
Patients satisfaction | 18 months
  Improvement of the scar assessed by the patient(Patient's global assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- The Netherlands Institute for Pigment Disorders, Amsterdam, Netherlands